CLINICAL TRIAL: NCT04884542
Title: A Prospective, Post-marketing Study Evaluating Clinical and Radiographic Early Outcomes of Revision Total Knee Arthroplasty With Multigen Plus H Alone or Involving AMF TT Cones.
Brief Title: Multigen Plus H Study and AMF TT Cones
Status: Recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Collaborators: North American Science Associates Ltd. (Network)
Responsible Party: Sponsor
Other Study IDs: K-23
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Revision Total Knee Arthroplasty — Total Knee Arthroplasty in case of failure of a previous operation.

SUMMARY:
The aim of this study is to assess the clinical, patient-reported, and radiographic outcomes of a revision Total Knee Arthroplasty with Multigen Plus H and AMF TT Cones.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥ 18 years old
* Given written informed consent approved by the reference Ethics Committee (EC)
* Subjects in whom a decision has already been made to perform a Total Knee Arthroplasty with the Multigen Plus H system as per Indication For Use. The decision to implant a Multigen Plus H system, alone or involving the AMF TT cones, must be taken prior to, and independently from, the decision to enrol the subject. This decision should be made in accordance with routine clinical practice at the study site concerned.
* Subject is able to comply with the protocol

Exclusion Criteria:

* Age < 18 years old
* Subjects with any Multigen Plus system contraindication for use, or any AMF TT cones contraindication for use when used in combination with the Multigen Plus H, as reported in the current Instruction For Use.
* Any clinically significant pathology based on the medical history or any medical intervention that the Investigator feels may affect the study evaluation
* Female subjects who are pregnant, nursing, or planning a pregnancy
* Previous knee replacement on the contralateral side within the last year and whose outcome is achieving an KSS < 70 points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population for this study includes adult subjects in whom the decision to perform a Total Knee Arthroplasty with Multigen Plus H system, alone or involving the AMF TT cones, must be taken prior to, and independently from, the decision to include the subject into the study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Knee Society Score (KSS) | Month 24
  Evaluation of the changes in the Functional Knee Society Score (KSS) after revision TKA

SECONDARY OUTCOMES:
KOOS-ADL (Function in Daily Living subdomain) | Month 24
  Evaluation of the functional changes in the KOOS-ADL domain after revision TKA
VAS Pain score | Month 24
  Evaluation of the changes in the VAS Pain score after revision TKA
Survivorship of the implant | Month 24
  Kaplan-Meier estimate
Radiographic implant evaluation and stability assessment | Month 24
  Evaluation of progressive Radiolucent Lines after revision TKA
Safety evaluation | Intra-operatively, Month 3, Month 12, and Month 24
  Incidence, type, and severity of all the Adverse Events (AEs) occurred after revision TKA

CONTACTS AND LOCATIONS:
Locations (2):
- AZ Jan Palfijn Gent, Ghent, Belgium
- Nemocnica Bory - Penta Hospital, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No